CLINICAL TRIAL: NCT00991380
Title: Healthy Eating & Active Living for Diabetes in Primary Care Networks
Acronym: HEALD-PCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alliance for Canadian Health Outcomes Research in Diabetes (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Jeffrey Johnson, Professor and Chair, The Alliance for Canadian Health Outcomes Research in Diabetes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Ach0rd-1001-09
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counselling (Experimental)
  Interventions: Behavioral: HEALD
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: HEALD — A six month, two phase pedometer-based walking program. For weeks one and two of phase I, participants will attend a group-based 60 minute education/supervised walking session. They will be asked to set a daily step goal and to attempt to achieve this on a daily basis over three months. Their steps will be recorded in a step log. For weeks one and two of phase II, participants will learn how to increase the speed of a portion of their daily steps and will learn the concept of low glycemic index and how to set dietary goals related to this concept. They will attend two sixty minute group-based education/supervised walking sessions.
  Other Names: Pedometer-based lifestyle intervention
  Arms: Lifestyle counselling
Behavioral: Usual Care — Control
  Other Names: Control, Usual care, off group
  Arms: Usual Care

SUMMARY:
The investigators aim to establish the effectiveness of a prescribed, community-based lifestyle modification program for those with recently diagnosed diabetes. The investigators hypothesize that those who enter a 6 month program will report greater levels of physical activity compared to a group who do not enter the program but who continue to receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* adult, recent type 2 diabetes diagnosis according to a diabetes patient registry, received a referral to a group-based lifestyle program or some provider-based diabetes related education.

Exclusion Criteria:

* physical limitation, cardiovascular contraindication, participation in any other research study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 3 months
Physical Activity | 6 months
Physical Activity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Johnson, PhD, Principal Investigator — University of Alberta; Steven T Johnson, PhD, Study Director — University of Alberta
Locations (1):
- The Alliance for Canadian Health Outcomes Research in Diabetes, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Johnson ST, Bell GJ, McCargar LJ, Welsh RS, Bell RC. Improved cardiovascular health following a progressive walking and dietary intervention for type 2 diabetes. Diabetes Obes Metab. 2009 Sep;11(9):836-43. doi: 10.1111/j.1463-1326.2009.01050.x. Epub 2009 Jul 10. PMID 19614943
- [Derived] Mathe N, Johnson ST, Wozniak LA, Majumdar SR, Johnson JA. Alternation as a form of allocation for quality improvement studies in primary healthcare settings: the on-off study design. Trials. 2015 Aug 25;16:375. doi: 10.1186/s13063-015-0904-x. PMID 26303892
- [Derived] Johnson ST, Mundt C, Soprovich A, Wozniak L, Plotnikoff RC, Johnson JA. Healthy eating and active living for diabetes in primary care networks (HEALD-PCN): rationale, design, and evaluation of a pragmatic controlled trial for adults with type 2 diabetes. BMC Public Health. 2012 Jun 19;12:455. doi: 10.1186/1471-2458-12-455. PMID 22712881
- See also: Click here for more details about the Alliance for Canadian Health Outcomes Research in Diabetes — http://www.achord.ca